CLINICAL TRIAL: NCT02138149
Title: Is the Nerve Growth Factor (NGF) a Useful Biomarker in Neurogenic Bladder Dysfunction After Spinal Cord Injury?
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2013-22
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Cord Injury; Neurogenic Detrusor Overactivity; Neurogenic Lower Urinary Tract Dysfunction
Keywords: spinal cord injury; neurogenic lower urinary tract dysfunction; nerve growth factor; neurogenic detrusor overactivity; urodynamics
MeSH Terms: conditions — Spinal Cord Injuries; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- spinal cord injury: individuals with neurogenic lower urinary tract dysfunction
- control group: individuals with physiologic bladder function

SUMMARY:
Spinal cord injury (SCI) almost always affects bladder function as well. As a result of this bladder dysfunction, individuals with SCI have to undergo regular invasive examination of their bladder function (urodynamic examination).

The nerve growth factor (NGF) is released from smooth muscle cells of the bladder, and there are reports, that the concentration of NGF is elevated in the urine of patients with bladder dysfunction. The NGF concentration can also be measured in the blood. The concentration of NGF in the blood and urine of SCI individuals has not yet been investigated. These concentrations may correlate with the severity of bladder dysfunction, and may thus be used to replace or at least reduce the number of the more invasive urodynamic examinations.

The hypothesis that urine and blood NGF concentrations in individuals with SCI are higher compared to individuals with healthy bladder function will be tested.

ELIGIBILITY:
Control Group

Inclusion Criteria:

* physiologic bladder function

Exclusion Criteria:

* no signed consent form
* age <18 / >80 years
* urinary tract infection
* bladder surgery
* radiation therapy of the pelvic area
* pregnancy
* bleeding disorder

Study Group

Inclusion Criteria:

* neurogenic detrusor overactivity
* presentation for urodynamic examination

Exclusion Criteria:

* no signed consent form
* age <18 / >80 years
* urinary tract infection
* bladder augmentation
* bladder evacuation by permanent catheterization
* radiation therapy of the pelvic area
* pregnancy
* bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals suffering from neurogenic lower urinary tract dysfunction, namely neurogenic detrusor overactivity
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
urinary concentration of nerve growth factor | day 0

SECONDARY OUTCOMES:
serum concentration of nerve growth factor | day 0
demographics | day 0
urodynamics | day 0
  only participants with spinal cord injury
International Prostate Symptom Score (I-PSS) | day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland